CLINICAL TRIAL: NCT02817126
Title: Robot-assisted Versus Laparoscopic Surgery for Mid/Low Rectal Cancer (REAL): A Multicenter Randomized Controlled Trial
Brief Title: Robot-assisted Versus Laparoscopic Surgery for Mid/Low Rectal Cancer
Acronym: REAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xu jianmin, Head of Colorectal Surgery, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REAL
Record Dates: First submitted 2016-03-07; First posted 2016-06-29 (Estimated); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Rectal Carcinoma
Keywords: Minimally Invasive Surgical Procedures; Robotic Surgical Procedures; Laparoscopic Surgical Procedures; Rectal Cancer; Intraoperative Complications; Postoperative Complications; Recovery of Function; Recurrence; Disease Progression; Survival
MeSH Terms: conditions — Rectal Neoplasms; Intraoperative Complications; Postoperative Complications; Recurrence; Disease Progression

ARMS (2):
- Robot-assisted surgery (Experimental): Patients undergo robot-assisted resections.
  Interventions: Procedure: Robot-assisted resection
- Laparoscopic surgery (Active Comparator): Patients undergo laparoscopic resections.
  Interventions: Procedure: Laparoscopic resection

INTERVENTIONS:
Procedure: Robot-assisted resection — Arm I: Robot-assisted resection using da vinci system.
  Arms: Robot-assisted surgery
Procedure: Laparoscopic resection — Arm II: Traditional laparoscopic resection.
  Arms: Laparoscopic surgery

SUMMARY:
The purpose of this study is to evaluate the safety and oncological feasibility of robot-assisted surgery for mid/low rectal carcinoma compared with laparoscopic surgery.

DETAILED DESCRIPTION:
Laparoscopic surgery as the treatment for colon cancer has been widely recognized. But its use for rectal cancer is still controversial. Previous trials have shown that although the long-term survival outcomes were similar, laparoscopic surgery did not reach the non-inferiority in terms of local tumor radical resection, compared with open surgery. Robotic techniques are considered to improve the quality of surgery with three-dimensional vision, stable camera platform and flexible robotic arms. Meta-analyses have shown that compared with laparoscopic surgery, robotic surgery could improve surgical quality in terms of open conversion, circumferential resection margin, postoperative complications, postoperative recovery, and quality of life, with similar long-term survival. However, these evidences mainly came from retrospective studies and small-scale randomized controlled trials with low quality. There still needs high-quality clinical trials to confirm the advantages of robotic surgery for rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) class I - III;
* Histologically proved rectal adenocarcinoma;
* Inferior tumor edge ≤ 10 cm from anal verge, measured by rigid rectoscopy;
* Tumor assessed as cT1-T3 (mesorectal fascia not involved) N0-1, or ycT1-T3 Nx after preoperative radio- or chemoradiotherapy, measured by pelvic MRI;
* No evidence of distant metastases;
* No other malignancies in medical history except adequately treated basocellular carcinoma of the skin or in situ carcinoma of the cervix uteri;
* Suitable for both robotic and laparoscopic surgery;
* Informed consent.

Exclusion Criteria:

* Tumors assessed as clinical complete response after preoperative radio- or chemoradiotherapy;
* Tumors assessed as cT1N0 and suitable for local excision;
* Signs of acute intestinal obstruction, bleeding or perforation needing emergency surgery;
* Multiple colorectal tumors or other schedules needing for synchronous colon surgery;
* Hereditary colorectal cancer (familial adenomatosis polyposis, Lynch Syndrome, etc.);
* Co-existent inflammatory bowel disease;
* Pregnancy or lactation;
* Patients received treatment other than preoperative radio- or chemoradiotherapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1240 (Actual)
Dates: Start 2016-07-10 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Locoregional recurrence rate | 3 years after surgery
  The proportion of patients with any cancer recurrence in the pelvic or perineal area

SECONDARY OUTCOMES:
Circumferential resection margin positive rate | 1 week after surgery
  The proportion of patients with circumferential resection margin ≤ 1 mm from the tumor
Postoperative complication rate | 30 days after surgery
  The proportion of patients with any complications occurred within 30 days after surgery
Overall survival time | 3 years after surgery
  Time from surgery to death
Disease-free survival time | 3 years after surgery
  Time from surgery to any recurrence, metastases or death
Operative time | Day 1
  Time from making skin incision to suturing the incision during the surgery
Rate of conversion to open surgery | Day 1
  The proportion of patients with the use of a laparotomy incision for any part of the TME procedure or lymph nodes dissection during the surgery
Estimated blood loss | Day 1
  Blood loss will be measured according to the suction and the weight of wet gauze, and then minus the irrigation.
Proximal/distal resection margin | 1 week after surgery
  The proximal/distal resection margin will be reported as "positive" or "negative" to define whether tumor is radically resected. It will be reported according to the post-operative pathology. Details are based on NCCN and Chinese guidelines for colorectal cancer.
Number of retrieved lymph nodes | 1 week after surgery
  The number of lymph node found from the surgical specimen
Postoperative hospital stay | 30 days after surgery
  The postoperative hospital stay is defined as the number of date from the first day after operation to discharge.
Self reported bladder function | At postoperative 3, 6 and 12 months
  This section is assessed using a self-rating scale "International prostate symptom score" (IPSS).
Self reported sexual function for male patients | At postoperative 3, 6 and 12 months
  This section is assessed using a self-rating scale "International Index of Erectile Function" (IIEF-5).
Self reported sexual function for female patients | At postoperative 3, 6 and 12 months
  This section is assessed using a self-rating scale "Female Sexual Function Index" (FSFI).

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Xu, Ph.D., M.D., Study Chair — Fudan University
Locations (11):
- China (11):
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - The Southwest Hospital of Army Medical University, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - Chinese PLA General Hospital of Northern Theatre Command (former Shenyang Military General Hospital), Shenyang, Liaoning
  - The 960th Hospital of Chinese PLA Joint Logistic Support Force (former Jinan Military General Hospital), Jinan, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Naval Medical University (Changhai Hospital), Shanghai, Shanghai Municipality

REFERENCES:
- [Derived] Feng Q, Yuan W, Li T, Tang B, Jia B, Zhou Y, Zhang W, Zhao R, Zhang C, Cheng L, Zhang X, Wei Y, Liang F, He G, Xu J; REAL Study Group. Robotic vs Laparoscopic Surgery for Middle and Low Rectal Cancer: The REAL Randomized Clinical Trial. JAMA. 2025 Jul 8;334(2):136-148. doi: 10.1001/jama.2025.8123. PMID 40455621
- [Derived] Feng Q, Yuan W, Li T, Tang B, Jia B, Zhou Y, Zhang W, Zhao R, Zhang C, Cheng L, Zhang X, Liang F, He G, Wei Y, Xu J; REAL Study Group. Robotic versus laparoscopic surgery for middle and low rectal cancer (REAL): short-term outcomes of a multicentre randomised controlled trial. Lancet Gastroenterol Hepatol. 2022 Nov;7(11):991-1004. doi: 10.1016/S2468-1253(22)00248-5. Epub 2022 Sep 8. PMID 36087608